CLINICAL TRIAL: NCT04095325
Title: Ultrasound Guided Transversus Abdominis Plane Block Versus Erector Spina Plane Block in Pediatric Lower Abdominal Surgery
Brief Title: Transversus Abdominis Plane Block Versus Erector Spina Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EBYU ESP
Record Dates: First submitted 2019-09-06; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Intraoperative Pain Control

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plane block (Active Comparator): Group 1 (n: 50): those who underwent TAP block after induction of propofol atropine and maintained with only 1 mg / kg / h propofol in anesthesia maintenance
  Interventions: Device: Ultrasound guided erector spinae block
- erector spinae block (Active Comparator): Group 2 (n: 50): those who underwent ESP block after propofol atropine induction and maintained with only 1 mg / kg / h propofol in anesthesia maintenance
  Interventions: Device: Ultrasound guided erector spinae block

INTERVENTIONS:
Device: Ultrasound guided erector spinae block — Group 2 (n: 50): those who underwent ESP block after propofol atropine induction and maintained with only 1 mg / kg / h propofol in anesthesia maintenance

SUMMARY:
Regional anesthesia and analgesia techniques are frequently used to provide pain control in pediatric surgical applications. The main advantages of these techniques include ease of application, good analgesic efficacy and low risk of complications (1). It reduces the need for parenteral opioids and increases the quality of postoperative pain control and the satisfaction of the patient and family (2). The aim of this study was to compare the contribution of TAP block and ESP block combined with sedation in pediatric surgery to anesthesia and analgesia during surgery without general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II,
* undergo elective lower abdominal surgery
* 2-6 years

Exclusion Criteria:

* Psychiatric patients,
* weight> 40 kg,
* those with cardiac-pulmonary-neurological disease,
* those with bleeding disorders,
* infection or wound scarring at the injection site,
* known allergy to local anesthetics

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 4 months
  effectiveness of erector spinae block on intraoperative anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kot P, Rodriguez P, Granell M, Cano B, Rovira L, Morales J, Broseta A, Andres J. The erector spinae plane block: a narrative review. Korean J Anesthesiol. 2019 Jun;72(3):209-220. doi: 10.4097/kja.d.19.00012. Epub 2019 Mar 19. PMID 30886130
- [Result] Tanaka M, Mori N, Murakami W, Tanaka N, Oku K, Hiramatsu R, Nakagawa M, Yasumoto K. [The effect of transversus abdominis plane block for pediatric patients receiving bone graft to the alveolar cleft]. Masui. 2010 Sep;59(9):1185-9. Japanese. PMID 20857679
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Hernandez MA, Palazzi L, Lapalma J, Cravero J. Erector spinae plane block for inguinal hernia repair in preterm infants. Paediatr Anaesth. 2018 Mar;28(3):298-299. doi: 10.1111/pan.13325. Epub 2018 Jan 17. PMID 29341379
- [Result] Stuart-Smith K. Hemiarthroplasty performed under transversus abdominis plane block in a patient with severe cardiorespiratory disease. Anaesthesia. 2013 Apr;68(4):417-20. doi: 10.1111/anae.12108. Epub 2012 Dec 17. PMID 23252578
- [Result] Tekelioglu UY, Demirhan A, Sit M, Kurt AD, Bilgi M, Kocoglu H. Colostomy with Transversus Abdominis Plane Block. Turk J Anaesthesiol Reanim. 2015 Dec;43(6):424-6. doi: 10.5152/TJAR.2015.89410. Epub 2015 Dec 1. PMID 27366540